CLINICAL TRIAL: NCT04187040
Title: SIMPLIFY the Hand Hygiene Procedure - Three Steps Versus Six Steps for Performing Hand Hygiene - an International Multicenter Cluster Randomized Trial (SIMPLIFY Study)
Brief Title: SIMPLIFY the Hand Hygiene Procedure - Three Steps Versus Six Steps for Performing Hand Hygiene (SIMPLIFY Study)
Acronym: SIMPLIFY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01071;me19Tschudinsutter2
Record Dates: First submitted 2019-11-12; First posted 2019-12-05 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hand Hygiene
Keywords: WHO-guideline on hand hygiene in healthcare; 3-step hand hygiene technique; 6-step hand hygiene technique

STUDY DESIGN:
Intervention Model Description: All participating wards will be randomly assigned with a 1:1 allocation to either the intervention (3-step hand hygiene technique) or the control group (6-step hand hygiene technique). Randomization will be stratified by participating institution for balanced allocation. Within each stratum, block randomization will be applied to assign wards to the two study groups. Blocking will be used to ensure close balance of the number of wards assigned to each group at any time during the study. Stratified randomization will be performed to ensure balance of the two groups within each institution.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-step hand hygiene technique (Active Comparator): Wards assigned to this study arm will receive instructions, educational materials and tutorials about the 3-step hand hygiene technique.
  Interventions: Procedure: Study intervention: 3-step hand hygiene technique
- 6-step hand hygiene technique (Active Comparator): Wards assigned to this study arm will receive instructions, educational materials and tutorials about the 6-step hand hygiene technique.
  Interventions: Procedure: Control intervention: 6-step hand hygiene technique

INTERVENTIONS:
Procedure: Study intervention: 3-step hand hygiene technique — 3-step hand hygiene technique:
  1. Covering all surfaces of the hands (based on own judgement)
  2. Rotational rubbing of fingertips in the palm of the alternate hand
  3. Rotational rubbing of both thumbs
  Arms: 3-step hand hygiene technique
Procedure: Control intervention: 6-step hand hygiene technique — 6-step hand hygiene technique (according to the WHO Guidelines on Hand Hygiene in Health Care, First Global Patient Safety Challenge):
  1. Rubbing hands palm to palm
  2. Palm to palm with fingers interlaced
  3. Right palm over left dorsum with interlaced fingers and vice versa
  4. Back of fingers to opposing palms with fingers interlocked
  5. Rotational rubbing of left thumb clasped in right palm and vice versa
  6. Rotational rubbing backwards and forwards with clasped fingers of right hand in left palm and vice versa
  Arms: 6-step hand hygiene technique

SUMMARY:
Hand hygiene is one of the most important measures to prevent healthcare associated infections. A hand hygiene technique consisting of three steps may be superior to the 6-step technique outlined by the World Health Organization (WHO) in terms of compliance with both indications and technique. Therefore, the aim of this study is to compare compliance with hand hygiene indications and technique between a 3-step and the 6-step technique for applying hand rub in an international multicenter cluster randomized trial.

DETAILED DESCRIPTION:
Hand hygiene is one of the most important measures to prevent transmission of pathogens between healthcare workers and patients, and ultimately, healthcare-associated infections. However, compliance with both hand hygiene indications and technique (outlining the steps for applying hand rub to ensure coverage of all surfaces of the hands) remains insufficient at most institutions worldwide. It was previously demonstrated that a hand hygiene technique consisting of three steps is superior to the 6-step technique outlined by the World Health Organization (WHO) in terms of compliance with both indications and technique in a single center study. Furthermore, the 3-step technique was non-inferior regarding microbiological efficacy in two experimental studies and during daily clinical practice. To further investigate the external validity and generalizability of these findings to different settings, this study compares both compliance with hand hygiene indications and technique between the 3-step and the 6-step technique for applying hand rub in an international multicenter cluster randomized trial.

ELIGIBILITY:
Inclusion Criteria:

Health Care Workers (HCW) working at the randomized wards during the pre-defined timeframe

Exclusion Criteria:

Individuals, who are no HCWs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compliance with hand hygiene indications | Up to one year
  Compliance with the five hand hygiene indications defined by the WHO:
  * before touching a patient
  * before clean/aseptic procedures
  * after body fluid exposure risk
  * after touching a patient
  * after touching patient surroundings
Compliance with the assigned hand hygiene technique | Up to one year
  Compliance with the assigned technique, defined as performance of the proposed three steps in the intervention group and of all six steps in the control group.

SECONDARY OUTCOMES:
Compliance with performance of the two steps for applying hand rub to the thumbs and the fingertips | Up to one year
  Compliance with performance of the two steps for applying hand rub to the thumbs and the fingertips, which are part of both the 3-step and the 6-step technique for applying hand rub.
Duration of the hand hygiene action | Up to one year
  Duration of the hand hygiene action, the time spent for the application of hand rub will be measured and compared between the two assignments.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin Sutter, Prof.Dr.med., Principal Investigator — University Hospital, Basel, Switzerland